CLINICAL TRIAL: NCT00337519
Title: Chemo-Immunotherapy With Allogeneic Blood Stem Cell Transplantation in Patients With Chronic Lymphocytic Leukemia (Study #02)
Brief Title: Allogeneic Stem Cell Transplantation in Chronic Lymphocytic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Hospital Carl Gustav Carus (Other); Deutsche Klinik fuer Diagnostik (Other)
Responsible Party: Dr. J. Schetelig, University Hospital Carl Gustav Carus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL #02; DJCLS-R03/01
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; reduced intensity conditioning; alemtuzumab; allogeneic stem cell transplantation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab

ARMS (1):
- 1 (Experimental): see detailed description
  Interventions: Procedure: allogeneic stem cell transplantation; Drug: Alemtuzumab

INTERVENTIONS:
Procedure: allogeneic stem cell transplantation — see detailed description
Drug: Alemtuzumab — alemtuzumab is given as cytoreductive pre-treatment with the last application of alemtuzumab scheduled for day 14

SUMMARY:
Patients with advanced chronic lymphocytic leukemia (CLL) have a poor long-term prognosis. Allogeneic stem cell transplantation (SCT) in patients with CLL has only rarely been performed in the past because the clinical outcome after myeloablative conditioning was poor, mainly due to the high treatment-related mortality. However long-term disease-free survival after allogeneic SCT has been reported. Recently it has been demonstrated by our group and others that non-relapse mortality can be reduced significantly with the use of reduced-intensity conditioning regimens. Yet, graft versus host disease (GVHD) remains an important problem in this setting.

Alemtuzumab is an effective drug for the treatment of patients with advanced CLL and has been successfully applied for GVHD-prophylaxis in the setting of myeloablative and reduced-intensity conditioning regimens. The goal of the present study is to evaluate the role of alemtuzumab as part of a fludarabine-based reduced intensity conditioning regimen for allogeneic SCT in patients with advanced CLL.

DETAILED DESCRIPTION:
Patients with relapsed or refractory CLL who are eligible for the study receive a cytoreductive therapy until SCT. Irrespective to the formal response, patients proceed to allogeneic SCT after fludarabine-based reduced-intensity conditioning. The use of granulocyte colony-stimulating factor (G-CSF)-mobilized peripheral blood stem cells > 3 x 10E6 CD34 cells/kg is recommended, but bone marrow > 1 x 10E8 MNC/kg is accepted. GVHD-prophylaxis is based on cyclosporine A adapted to blood levels (150 to 200 ng/mL) over a period of three months. In Phase I of the study, alemtuzumab has been applied as part of the conditioning regimen until day 5. In Phase II, alemtuzumab is given as cytoreductive pre-treatment with the last application of alemtuzumab scheduled for day 14 and after Amendment II in September 2006 scheduled for day 28. Furthermore methotrexate is given on days 1, 3, 6. and 11 at a projected cumulative dose of 45 mg/m2. Subsequent immunosuppressive therapy depends on the occurrence of GvHD, the development of chimerism, and residual disease. Patients with relapsing or residual disease (minimal residual disease excluded) who do not suffer from GvHD should receive donor lymphocytes in increasing dosages. The initial dose is 1 x 105/kg T-cells in unrelated donors and 1 x 106/kg in matched related donors. If no GvHD develops within 6-8 weeks, the next higher dosage is applied.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* sufficient organ function
* availability of an HLA-compatible donor (related or unrelated)
* age < 65 years
* karnofsky index > = 70%
* B-CLL requiring treatment after failure of at least one prior cytostatic treatment

Exclusion Criteria:

* positive HIV-serology
* pregnancy
* intolerance to study drugs
* second neoplasia
* serious infections

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2003-01; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 400 days

SECONDARY OUTCOMES:
safety according to common toxicity criteria (CTC) | at discharge and until last follow up
rate of primary and secondary graft failure | until last follow up
rate of acute and chronic GVHD | day 100 and last follow up
response rate | 2 years
chimerism | day 100

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schetelig, MD, Study Chair — University Hospital Carl Gustav Carus, Dresden
Locations (3):
- Germany (3):
  - Klinikum Chemnitz gGmbH, Chemnitz, Chemnitz
  - Uniklinikum Carl Gustav Carus, Dresden
  - Deutsche Klinik für Diagnostik GmbH, Wiesbaden